CLINICAL TRIAL: NCT01718886
Title: Feasibility Study to Evaluate Preliminary Safety and Efficacy of Multiple Obalon Gastric Balloons for 12 Weeks as an Aid for Weight Loss
Brief Title: European Study to Evaluate Preliminary Safety and Efficacy of Multiple Obalon Gastric Balloons for 12 Weeks as an Aid for Weight Loss
Status: Completed | Type: Observational
Sponsor: Obalon Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PTL-1000-0018
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Obesity; Weight Control
Keywords: Obesity; Weight loss; Weight control; Intragastric balloon; gastric balloon
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Obalon Gastric Balloon: Patients received 1-3 Obalon Gastric Balloons over a period of 12 weeks
  Interventions: Device: Obalon Gastric Balloon

INTERVENTIONS:
Device: Obalon Gastric Balloon

SUMMARY:
The objective of this study is to evaluate the initial safety and preliminary effectiveness of the Obalon intragastric balloon system in European subjects with a BMI in the range of 27 - 35 kg/m^2

ELIGIBILITY:
Inclusion Criteria:

* Were between 21-64 years of age;
* Had a BMI 27-35 Kg/cm
* Did not have a history of weight reduction over 5% of body weight over the past 6 months
* Were able to comply with all study requirements for the duration of the study as outlined in the protocol. This included complying with the visit schedule as well as study specific procedures such as: electrocardiography, endoscopy, upper gastrointestinal radiography and clinical lab testing
* Were able to understand and willing to provide written informed consent

Exclusion Criteria:

* Experienced any difficulty in swallowing;
* Had unstable angina, myocardial infarction within the past year, or heart disease classified within the New York Heart Association's Class III or IV functional capacity;
* Taking chronic aspirin or other non steroidal anti-inflammatory agents, or other medications known to be gastric irritants, and not willingness to discontinue the use of these concomitant medications, antiarrythmics, anti-anginal medications, anticoagulants or medications for congestive heart failure;
* Taking blood pressure medications, unless their blood pressure was controlled and they have been at stable dose for at least 3 months;
* Had type 1 diabetes or Type 2 diabetes requiring oral medications or insulin;
* Had a history or symptoms of thyroid disease which is not controlled by medication;
* Had severe renal, hepatic, pulmonary disease or cancer;
* Had past history of gastrointestinal surgery (excluding uncomplicated appendectomy);
* Had any abnormal stenosis or obstruction of the GI tract;
* Had a history of adhesive peritonitis;
* Had a previously diagnosed hiatal hernia greater than 2cm;
* Had any abnormality of the esophagus, stomach or pylorus;
* Had history of severe esophagitis;
* Had history or symptoms of esophageal and/or gastric varices;
* Had history or congenital or acquired GI anomalies (e.g. atresias, stricture, and /or diverticula);
* Had history or symptoms of inflammatory bowel disease, such as Chron's disease;
* Had history of/ signs and /or symptoms of duodenal or gastric ulcer;
* Untreated H.Pylori
* Had history or signs of dysphasia, achalasia or symptoms of or GI motility;
* Were undergoing chronic steroid or immunosuppressive therapy;
* Were pregnant or breastfeeding or had the intention of becoming pregnant during the study;
* Had placement of previous intragastric balloon or similar device;
* Were using pharmaceutical agents for weight loss;
* Were drinking alcohol in excess or using illicit drugs;
* Had bulimia or binge eating disorders;
* Had impending gastric surgery 30 days post balloon removal;
* Had planned flying or scuba diving activities during balloon residence time;
* Had any other condition that, in the opinion of the investigator, would interfere with their participation and compliance with the study (i.e. psychosocial issues);
* Were participating in other investigational study protocols. If a subject had recently completed participation in another drug or device study, the subject must have completed that study at least 30 days prior to being enrolled in this study;
* Had history or known allergies to any component of the device materials, including but not limited to allergies to porcine proteins.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients were selected from investigators' patient population and included patients with a BMI in the range of 27 - 35 kg/m^2
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Percent Excess Weight Loss based on an ideal BMI of 25. | 12 weeks
Assessment of all adverse events. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fancois Mion, MD, Principal Investigator — Hospital Edouard Harriot; Jacques Deviere, Principal Investigator — Erasme University Hospital
Locations (2):
- Department of Gastroenterology, Erasme Hospital, Brussels, Belgium
- Service D'exploration Functionelle Digestive, Hospital Edouard Harriot, Lyon, Cedex, France

REFERENCES:
- See also: Sponsor's website — http://www.obalon.com